CLINICAL TRIAL: NCT06412224
Title: An Exploratory ITT（Investigator Initiated Study) Study to Evaluate the Preliminary Safety and Efficacy of Single Subretinal Injection of RRG001 at the End of or After Vitrectomy in Subjects With PDR
Brief Title: The Preliminary Safety and Efficacy of RRG001 After Vitrectomy in Subjects With Proliferative Diabetic Retinopathy (PDR)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Li Xiaorong (Other)
Collaborators: Shanghai Refreshgene Technology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Li Xiaorong, Assistant Investigator, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRG001-P01
Record Dates: First submitted 2024-04-24; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: PDR - Proliferative Diabetic Retinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RRG001 (Experimental): Frequency of administration: one time injection.
  Interventions: Drug: RRG001

INTERVENTIONS:
Drug: RRG001 — Administered by subretinal injection. Dosage form: injection.

SUMMARY:
This study aims to slow down disease progression, reduce postoperative complications and decrease retreatment frequency in subjects with proliferative diabetic retinopathy (PDR) by administering a single subretinal injection of RRG001 gene therapy after vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Age >= 20 years
* Diagnosis of diabetes mellitus (type 1 or type 2)
* The study eye diagnosed with PDR, in the opinion of the investigator, requires vitrectomy and postoperative anti-VEGF therapy, or that has undergone vitrectomy and still requires postoperative anti-VEGF therapy
* Based on the ETDRS chart, the best-corrected visual acuity (BCVA) of the study eye is ≥ hand motion and ≤ 63 letters

Exclusion Criteria:

* Active infection or inflammation in either eye
* Previous gene therapy in either eye
* Uncontrolled blood pressure（defined as systolic ≥160mmHg or diastolic ≥ 110mmHg by anti-hypertensive treatment)
* HbA1c >12% for diabetes patients at screening
* Previous condition not eligible for study drug
* History of major ocular surgery (except for PDR) or severe trauma
* Currently enrolled in another clinical trial or planning to enroll during the study
* Pregnant or lactating women
* Other conditions that, in the opinion of the investigator, would preclude participation in the study

Study Eye-Exclusion Criteria：

* Ocular disorders that, in the opinion of the investigator, would confound the interpretation of study results or affect the administration
* CNV or macular edema secondary to any causes other than diabetic retinopathy
* Ocular condition considered by the investigator to contraindicate subretinal injection
* Diagnosed primary or secondary glaucoma
* History of intraocular corticosteroid treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of DLTs (dose limiting toxicity analysis) at most 6 subjcts | Within 28 days after RRG001 administration
  To evaluate the incidence of DLTs (dose limiting toxicity analysis) at most 6 subjcts
To evaluate the incidence of AEs(Adverse Event) as assessed CTCAE 5.0 at most 6 subjcts | Within 24 weeks after RRG001 administration
  To evaluate the incidence of AEs as assessed CTCAE 5.0 at most 6 subjcts

SECONDARY OUTCOMES:
To evaluate the disease progression as assessed the vitreous hemorrhage of the study eye at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the disease progression as assessed the vitreous hemorrhage of the study eye at most 6 subjects
To evaluate the disease progression as assessed the retinal detachment of the study eye at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the disease progression as assessed the retinal detachment of the study eye at most 6 subjects
To evaluate the frequency for rescue therapy of the study eye at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the frequency for rescue therapy of the study eye at most 6 subjects
To evaluate the change from baseline in BCVA(Best Corrected Visual Acuity) of the study eye as assessed by ETDRS chart at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the change from baseline in BCVA of the study eye as assessed by ETDRS chart at most 6 subjects
To evaluate the anatomical changes of the study eye by OCT(optical coherence tomography) at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the anatomical changes of the study eye by OCT(optical coherence tomography) at most 6 subjects
To evaluate the anatomical changes of the study eye by CFP(colour fundus photography）at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the anatomical changes of the study eye by CFP(colour fundus photography）at most 6 subjects
To evaluate the anatomical changes of the study eye by OCTA（optical coherence tomography angiography) at most 6 subjects | Within 24 weeks after RRG001 administration
  To evaluate the anatomical changes of the study eye by OCTA（optical coherence tomography angiography) at most 6 subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No